CLINICAL TRIAL: NCT00392782
Title: A Multicenter, Prospective Trial to Evaluate the Role of NK Cell KIR Epitope Mismatch on Mortality and Disease Relapse in T-Cell Depleted Hematopoietic Stem Cell Transplantation From HLA-C Mismatched, Unrelated Donors for Myeloid Malignancies
Brief Title: Donor Stem Cell Transplant in Treating Patients With Myeloid Cancer or Other Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Center for International Blood and Marrow Transplant Research (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004UC035; UMN-MT2004-04 (Other: Blood and Marrow Transplantation Program); UMN-0405M59662 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Results first posted 2011-07-15 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia in remission; childhood acute myeloid leukemia in remission; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; secondary myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Accelerated Phase; Blast Crisis | interventions — Antilymphocyte Serum; fludarabine phosphate; Thiotepa; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Natural Killer Cell Kir Epitope (Experimental)
  Interventions: Biological: anti-thymocyte globulin; Drug: fludarabine phosphate; Drug: thiotepa; Procedure: peripheral blood stem cell transplantation; Radiation: total-body irradiation

INTERVENTIONS:
Biological: anti-thymocyte globulin — Rabbit thymoglobulin will be given intravenously at a dose of 2.5 mg/kg on days -5,-4, -3, and -2. The first dose of thymoglobulin will be given over six (6) hours and subsequent doses over four (4) or more hours as tolerated or, per institutional anti-thymocyte globulin (ATG) administration guidelines.
  Other Names: ATG
Drug: fludarabine phosphate — Fludarabine 40 mg/m^2/day intravenously (IV) over 30-60 minutes on days -7,-6,-5,-4,-3 (total dose 200 mg/m^2).
  Other Names: Fludara
Drug: thiotepa — Thiotepa 5 mg/kg/day intravenously (IV) over 4 hours on days -8, -7 (total dose 10 mg/kg).
Procedure: peripheral blood stem cell transplantation — Peripheral Blood Stem Cell (PBSC) Infusion. All patients will receive granulocyte colony-stimulating factor (G-CSF)-mobilized PBSC on day 0 (or day+1 when available) following CD34 cell selection for ex vivo T cell removal. PBSC is infused via a central venous catheter using blood infusion tubing.
  Other Names: PBSC
Radiation: total-body irradiation — The total-body irradiation (TBI) will be given in 2 fractions of 400 cGy each administered on day -10 and -9 via anterior and posterior fields for a total dose of 800 cGy.
  Other Names: TBI

SUMMARY:
RATIONALE: Giving total-body irradiation and chemotherapy, such as fludarabine and thiotepa, before a donor stem cell transplant helps stop the growth of cancer or abnormal cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When healthy stem cells from a donor are infused into the patient, they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving antithymocyte globulin and removing the T cells from the donor cells before transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well a donor stem cell transplant works in treating patients with myeloid cancer or other disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the incidence of disease-free survival at 1 year in patients with acute or chronic myeloid leukemias undergoing T-cell-depleted hematopoietic stem cell transplantation from HLA-C mismatched, unrelated donors.

Secondary

* Determine the incidence of disease relapse at 1 year in patients treated with this regimen.
* Determine the incidence and severity of acute graft-vs-host disease (GVHD) at 100 days and chronic GVHD at 1 year in these patients.
* Determine the incidence of graft failure at day 100.
* Determine the transplant-related mortality of these patients at 1 year.
* Determine the overall survival of these patients at 1 year.

OUTLINE: This is a prospective, multicenter study. Patients are stratified according to killer-cell immunoglobulin-like receptors (KIR) epitope mismatch (yes [experimental] vs no [control]).

* Myeloablative preparative regimen: Patients undergo total body irradiation twice daily on days -10 and -9 and receive thiotepa intravenously (IV) over 4 hours on days -8 and -7, fludarabine phosphate IV over 30-60 minutes on days -7 to -3, and antithymocyte globulin IV over 4-6 hours on days -5 to -2.
* Allogeneic peripheral blood stem cell (PBSC) transplantation: Patients undergo filgrastim (G-CSF)-mobilized, T-cell-depleted, CD34+-selected allogeneic PBSC transplantation on day 0.

After completion of study treatment, patients are followed periodically for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Primary acute myeloid leukemia (AML)

  * First complete remission (CR) with high risk features as defined by: failure to achieve remission by day 21 after induction chemotherapy, or the presence of chromosomal abnormalities involving any of the following: -5/de (5q), -7/del(7q), inversion 3q, abnormalities of 11q23, 20q, 21q, del(9q), translocation 6;9, translocation 9;22, abnormalities of 17p, or complex karyotype with > or = 3 abnormalities. Complete remission is defined as < 5% blasts in the marrow.
  * Second CR or subsequent in remission
  * Refractory or relapsed disease with absolute peripheral blood blasts < 2000/mcL
* Secondary AML in remission or relapse
* Chronic myelogenous leukemia (CML) in accelerated or blast phase

  * Accelerated phase is defined by any one of the following:

    * Blasts 10% to 19% of peripheral blood white cells or bone marrow cells
    * Peripheral blood basophils at least 20%
    * Persistent thrombocytopenia (<100 x 10^9/L) unrelated to therapy, or persistent thrombocytosis (>1000 x 10^9/L) unresponsive to therapy
    * Increasing spleen size and increasing white blood cell (WBC) count unresponsive to therapy
    * Cytogenetic evidence of clonal evolution (i.e., the appearance of an additional genetic abnormality that was not present in the initial specimen at the time of diagnosis of chronic phase CML)
    * Resistance to tyrosine kinase inhibitors (imatinib or other) defined as no complete cytogenetic response even if the above criteria are not met.
  * Blast phase is defined by either of the following:

    * Blasts 20% or more of peripheral blood white cells or bone marrow cells
    * Extramedullary blast proliferation
    * Large foci or clusters of blasts in bone marrow biopsy
* Primary myelodysplastic syndrome (MDS) with an IPSS score >1
* Secondary MDS with any international prostate symptom score (IPSS)
* Age ≤60 years
* Co-Morbidity score 0-2
* At least 35 days following start of preceding leukemia induction therapy

Exclusion Criteria:

* Patients for whom a suitable HLA genotypically identical sibling or fully matched HLA-A, -B, -C, and -DRB1 unrelated donor is available.
* Patients greater than 60 years of age.
* Hypersensitivity to thymoglobulin.
* Symptomatic uncontrolled coronary artery disease or congestive heart failure.
* Hepatic disease with transaminases or bilirubin > 2 times upper limit of normal (ULN) except for isolated hyperbilirubinemia attributed to Gilbert's syndrome.
* Severe hypoxemia with room air - Partial Pressure of Oxygen in Arterial Blood - (PAO2) < 70, supplemental oxygen-dependence, or carbon monoxide diffusing capacity (DLCO) < 50% predicted.
* Impaired renal function with creatinine > 2 times upper limit of normal (ULN) or creatinine clearance measured by 24-hour urine collection < 50% normal for age, gender, and weight.
* Patients with central nervous system (CNS) involvement with disease refractory to intrathecal chemotherapy.
* Patients who are human immunodeficiency virus (HIV) seropositive.
* Patients who are pregnant or breast-feeding.
* Patients with active infections that are untreated, or failing to respond to appropriate therapy.
* Karnofsky performance status < 50%.
* Prior allogeneic or autologous bone marrow, peripheral blood stem cell, or umbilical cord blood transplant.
* Inability to provide informed consent.
* Co-morbidity score >2
* Less than 35 days from start of previous leukemia induction therapy

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2005-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Weisdorf, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (9):
- United States (9):
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Midwest Children's Cancer Center at Children's Hospital of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- All Treated Patients: Includes patients with partial matched unrelated donor transplants and treated with: total body irradiation twice daily on days -10 and -9 and receive thiotepa intravenously (IV) over 4 hours on days -8 and -7, fludarabine phosphate IV over 30-60 minutes on days -7 to -3, and antithymocyte globulin IV over 4-6 hours on days -5 to -2.
  Patients undergo filgrastim (G-CSF)-mobilized, T-cell-depleted, CD34+-selected allogeneic PBSC transplantation on day 0.
Period: Overall Study
Arm/Group | All Treated Patients
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Treated Patients
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
Disease [Number; unit: Participants]
  Acute Myeloid Leukemia - CR1 | 10
  Acute Myeloid Leukemia - CR2 | 7
  Myelodysplastic Syndrome - RAEB2 | 2
  Myelodysplastic Syndrome - NOS | 1
  Chronic Myeloid Leukemia | 4

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Disease-free Survival
Description: Number of patients alive and without disease at 1 year after transplant.
Time Frame: 1 Year
Measure: Number; unit: Participants
Arm/Group | All Treated Patients
Number analyzed (Participants) | 24
Participants | 18

2. Secondary Outcome: Incidence of Disease Relapse
Description: Number of patients with disease at 1 year.
Time Frame: 1 Year
Measure: Number; unit: Participants
Arm/Group | All Treated Patients
Number analyzed (Participants) | 24
Participants | 6

3. Secondary Outcome: Incidence of Grade II-IV Acute Graft-vs-host Disease (GVHD)
Description: Number of patients with grade II-IV acute graft-versus-host disease at Day 100 post transplant. Graft-versus-host disease (GVHD) is a common complication of allogeneic bone marrow transplantation in which functional immune cells in the transplanted marrow recognize the recipient as "foreign" and mount an immunologic attack. Grade I=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life threatening.
Time Frame: Day 100
Measure: Number; unit: Participants
Arm/Group | All Treated Patients
Number analyzed (Participants) | 24
Participants | 6

4. Secondary Outcome: Incidence of Chronic Graft-versus-host Disease (GVHD)
Description: Number of patients with chronic graft-versus-host disease at 1 year post transplant. Graft-versus-host disease (GVHD) is a common complication of allogeneic bone marrow transplantation in which functional immune cells in the transplanted marrow recognize the recipient as "foreign" and mount an immunologic attack. Grade I=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life threatening. Chronic GVHD is an extension of acute GVHD.
Time Frame: 1 Year
Measure: Number; unit: Participants
Arm/Group | All Treated Patients
Number analyzed (Participants) | 24
Participants | 4

5. Secondary Outcome: Incidence of Graft Failure
Description: Number of patients with graft failure is defined by lack of neutrophil engraftment by 100 days after transplant in patients surviving a minimum of 14 days.
Time Frame: Day 100
Measure: Number; unit: Participants
Arm/Group | All Treated Patients
Number analyzed (Participants) | 24
Participants | 1

6. Secondary Outcome: Transplant-related Mortality
Description: Number of patients with treatment related death at 1 year post transplant.
Time Frame: 1 Year
Measure: Number; unit: Participants
Arm/Group | All Treated Patients
Number analyzed (Participants) | 24
Participants | 8

7. Secondary Outcome: Overall Survival
Description: Number of patients who were deceased at 1 year post transplant.
Time Frame: 1 Year
Measure: Number; unit: Participants
Arm/Group | All Treated Patients
Number analyzed (Participants) | 24
Participants | 10

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from first date of study treatment up to 1 year post transplant.
Description: Because all study participants received potentially toxic preparative therapy, significant regimen-related toxicity was anticipated. Therefore only selected adverse events (serious infections, graft failure and GVHD) were collected.
Arm/Group | All Treated Patients
Serious Adverse Events (participants affected / at risk) | 23/24
Other Adverse Events (participants affected / at risk) | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Patients (N=24)
ALT/serum glutamic pyruvic transaminase increased (Immune system disorders) | 1 (1)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1)
Blood/bone marrow, other (Blood and lymphatic system disorders) | 2 (2)
Cerebrovascular ischemia (Nervous system disorders) | 1 (1)
Cardiac, general (Cardiac disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Death (General disorders) | 3 (3)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Low serum glucose (Endocrine disorders) | 1 (1)
Low hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection with Grade 3-4 neutrophils (Blood and lymphatic system disorders) | 1 (2)
Infection, other (Infections and infestations) | 3 (4)
Infection with normal neutrophils, lung (Infections and infestations) | 1 (2)
Infection with unknown neutrophils, blood (Infections and infestations) | 6 (6)
Infection with unknown neutrophils, catheter (Infections and infestations) | 2 (2)
Infection with unknown neutrophils, colon (Infections and infestations) | 1 (1)
Infection w/unknown neutrophils - lung (Infections and infestations) | 1 (1)
Infection w/unknown neutrophils - mucosa (Infections and infestations) | 1 (1)
Infection with unknown neutrophils - upper airway (Infections and infestations) | 1 (1)
Infection with unknown neutrophils - wound (Infections and infestations) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal necrosis (General disorders) | 1 (1)
Neurology (Nervous system disorders) | 1 (2)
Gastrointestinal obstruction - ureter (Gastrointestinal disorders) | 1 (1)
Pain - abdomen (General disorders) | 2 (2)
Pain - cardiac/heart (Cardiac disorders) | 1 (1)
Progressive disease (General disorders) | 1 (1)
Pulmonary - upper respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Relapse (General disorders) | 2 (2)
Renal (Renal and urinary disorders) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thrombosis (Blood and lymphatic system disorders) | 2 (2)
Vascular (Cardiac disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes